CLINICAL TRIAL: NCT01410396
Title: Occult Paroxysmal Atrial Fibrillation in Patients With Non-cardioembolic Ischemic Stroke of Determined Mechanism
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: LifeWatch Services, Inc. (Industry)
Responsible Party: Principal Investigator, Richard Bernstein, Associate Professor, Stroke/Cerebrovascular, Northwestern University
Other Study IDs: Lifewatch
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the yield of 3 weeks outpatient mobile cardiac monitoring for detection of atrial fibrillation in patients with history of stroke of known cause.

DETAILED DESCRIPTION:
Patients will be recruited to wear a outpatient mobile cardiac monitoring device for detection of atrial fibrillation in patients with a history of stroke of known case. Their are not study treatments or interventions, this is an observational trial. Eligible patients must be >50 years old, have a history of ischemic stroke or transient ischemic attack with a documented brain infarction within the prior 12 months. If patients are on anticoagulation therapies, they are eligible for enrollment if the long-term strategy for stroke prevention is anti-platelet therapy and not the oral anti-coagulant itself. Patients must not have an detection of AF and then must successfully activate the lifeStar device for enrollment. At the end of three weeks, the LifeStar device will be over-read and scored for the presence of AF and other clinically significant arrhythmias by the study electrophysiologist, who will determine the occurrence and burden of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50
2. Ischemic stroke, or transient ischemic attack with documented acute brain infarction, within prior 6 months.
3. Patient does not merit indefinite oral anticoagulation. (Patients requiring temporary OAC for purposes other than recurrent stroke prevention, such as treatment of a deep venous thrombosis, are eligible for enrollment if the long-term secondary stroke preventive strategy is anti-platelet therapy and not OAC).
4. Stroke mechanism is determined to be lacunar stroke, large vessel intracranial atherosclerosis, large vessel extracranial atherosclerosis, or a combination thereof.
5. Patient has been evaluated with at least a 12 lead EKG and at least one day of in-patient or out-patient cardiac telemetry, with no detection of AF or atrial flutter.
6. Detection of AF or atrial flutter would change secondary prevention antithrombotic strategy (eg to indefinite OAC).
7. Patient receives and successfully activates LifeStar ACT device.
8. Patient or legally authorized representative signs informed consent.

Exclusion Criteria:

1. Known history of AF or atrial flutter.
2. Patient has defibrillator or pacemaker capable of detecting AF.
3. Patient has indication for indefinite OAC.
4. Patient has indefinite contra-indication to OAC. (Patients with temporary ineligibility for OAC, for example due to the need for invasive medical procedures or large acute brain infarction, are eligible for enrollment).
5. Stroke due to known cause not listed in inclusion criterion 4.
6. Cardioembolic stroke.
7. Inability to comply with LifeStar ACT monitoring regimen.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of stroke of known mechanism age greater than 50
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Detection of any episode of AF >30 seconds during 21 days of mobile outpatient cardiac telemetry | 21 days

SECONDARY OUTCOMES:
Recurrent ischemic stroke | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bernstein, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States